CLINICAL TRIAL: NCT04126902
Title: Analyses of Interleukin-6, Presepsin and Pentraxin-3 in the Diagnosis and Severity of Late-onset Preeclampsia
Acronym: Presepsin&PE
Status: Completed | Type: Observational
Sponsor: Cengiz Gokcek Women's and Children's Hospital (Other)
Responsible Party: Principal Investigator, Ali Ovayolu, Principal Investigator, Cengiz Gokcek Women's and Children's Hospital
Other Study IDs: CengizGWCH5
Record Dates: First submitted 2019-10-10; First posted 2019-10-15 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Preeclampsia
Keywords: innate immunity; macrophage; toll-like receptors; trophoblasts; phagocytos
MeSH Terms: conditions — Pre-Eclampsia | interventions — Interleukin-6; PTX3 protein

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- late-onset preeclampsia: The diagnosis of L-PrE, as defined by the Committee on Terminology of the American College of Obstetricians and Gynecologists (ACOG), is established based on the presence of proteinuria (urinary excretion of protein ≥300 mg in a 24-h urine specimen, or proteinüria ≥1+ in dipstick) and a blood pressure level of ≥90/140 mmHg (two blood pressure measurements 6 h apart) that occurs after 34 weeks of gestation in a previously normotensive woman. The diastolic and/or systolic blood pressure <110/160 mm Hg, it was accepted as mild; and in case these values exceeded this level, it was accepted as severe. The study population consisted of 50 late-onset preeclampsia patients as study group and 50 patients with normal pregnancies as control group.
  Interventions: Other: interleukin-6, presepsin and pentraxin-3
- Control: The control groups' samples obtained during the routine obstetrical care examination in the third trimester of pregnancy. Then these pregnant women followed-up until the delivery.
  Interventions: Other: interleukin-6, presepsin and pentraxin-3

INTERVENTIONS:
Other: interleukin-6, presepsin and pentraxin-3 — measurements and compare

SUMMARY:
Introduction: The etiology/pathophysiology of preeclampsia remains an enigma. Cellular immunity is a key factor in the etiology of late-onset preeclampsia (L-PrE). Presepsin is split out from the phagocytes membranes after phagocytosis. To investigators knowledge, this is the first study in literature to investigate maternal blood concentrations of presepsin in preeclampsia and healthy pregnant women.

Methods: The investigators examined maternal plasma interleukin-6, presepsin and pentraxin-3 concentrations in pregnant women with (n=44) and without L-PrE (n=44). These three inflammatory markers concentrations measured using enzyme-linked immunosorbent assays were compared.

DETAILED DESCRIPTION:
This observational case-control study was designed at Cengiz Gokcek Women's and Children's Hospital, Gaziantep, Turkey, in the Department of Obstetrics and Gynecology between June 2018 and January 2019. The protocol was approved by the Ethics Committee for Clinical Research of Gaziantep University (Reference number: 2018/393). The study strictly adhered to the principles of the Declaration of Helsinki. All subjects included in the study gave oral and written informed consent. Eighty-eight women were enrolled in the study in two groups. All participants will gave their oral and written informed consent before their inclusion in the study.

ELIGIBILITY:
Inclusion Criteria:

* preeclampsia healthy pregnancy

Exclusion Criteria:

1. pregnant women with any systemic condition (such as chronic hypertension, inflammatory and rheumatic diseases),
2. using any kind of medication throughout pregnancy (such as acetylsalicylic acid, corticosteroids or heparin),
3. pregnant women who had fever at the time of the first admission,
4. concurrent infections (urinary tract infection, cervicitis, etc.),
5. pregnancies complicated with premature membrane rupture or chorioamnionitis,
6. history of medication for PE treatment at the time of the first admission,
7. patients who had fetal congenital abnormalities or genetic syndromes,
8. drug user,
9. multiple gestations,
10. active labor.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnancy- preeclampsia
Study Population: The investigators consecutively recruited 50 subjects with preeclampsia, and 50 healthy pregnancies selected for the control group.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
The primary endpoint in these analyses was IL-6, presepsin and pentraxin-3 levels in late-onset preeclampsia group and control group. | 3 months
  The primary endpoint in these analyses was IL-6, presepsin and pentraxin-3 levels in late-onset preeclampsia and control group.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ovayolu, MD, Principal Investigator — Cengiz Gokcek WCH
Locations (1):
- Cengiz Gokcek Women's and Child's hospital, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Magee LA, Pels A, Helewa M, Rey E, von Dadelszen P; Canadian Hypertensive Disorders of Pregnancy (HDP) Working Group. Diagnosis, evaluation, and management of the hypertensive disorders of pregnancy. Pregnancy Hypertens. 2014 Apr;4(2):105-45. doi: 10.1016/j.preghy.2014.01.003. Epub 2014 Feb 25. PMID 26104418
- [Background] Hypertension in pregnancy. Report of the American College of Obstetricians and Gynecologists' Task Force on Hypertension in Pregnancy. Obstet Gynecol. 2013 Nov;122(5):1122-1131. doi: 10.1097/01.AOG.0000437382.03963.88. No abstract available. PMID 24150027
- [Result] Canzoneri BJ, Lewis DF, Groome L, Wang Y. Increased neutrophil numbers account for leukocytosis in women with preeclampsia. Am J Perinatol. 2009 Nov;26(10):729-32. doi: 10.1055/s-0029-1223285. Epub 2009 May 18. PMID 19452432
- [Result] Pugni L, Pietrasanta C, Milani S, Vener C, Ronchi A, Falbo M, Arghittu M, Mosca F. Presepsin (Soluble CD14 Subtype): Reference Ranges of a New Sepsis Marker in Term and Preterm Neonates. PLoS One. 2015 Dec 31;10(12):e0146020. doi: 10.1371/journal.pone.0146020. eCollection 2015. PMID 26720209

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-10): https://cdn.clinicaltrials.gov/large-docs/02/NCT04126902/Prot_SAP_000.pdf